CLINICAL TRIAL: NCT01162135
Title: A Pilot Phase II Study of Digoxin in Patients With Recurrent Prostate Cancer as Evident by a Rising PSA
Brief Title: Digoxin for Recurrent Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10G.87; 2009-43 (Other: CCRRC); JT 1532 (Other: JeffTrial Number)
Record Dates: First submitted 2010-07-12; First posted 2010-07-14 (Estimated); Results first posted 2014-06-05 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Digoxin; Recurrent Prostate Cancer; Prostate Specific Antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label Pilot Study (Experimental)
  Interventions: Drug: Digoxin

INTERVENTIONS:
Drug: Digoxin — The participants will take study drug digoxin, which is approved by FDA for the treatment of CHF, 125 or 250 mcg orally daily, titrated to the level of 0.8 - 2 ng/ml for total of 6 cycles (4 weeks/cycle). The lower dose of digoxin (such as 125 mcg/day) will be chosen if serum level reaches 0.8 ng/ml already. Patients may continue another 6 cycles if evident of clinical benefit.
  It is possible that some patients may need to receive 500 mcg per day to reach this targeted drug level. No further titration will be allowed beyond this FDA approved digoxin dose.

SUMMARY:
The purpose of this study is to assess the effectiveness of dioxin on prohibiting prostate cancer progression as measured by PSADT (prostate-specific antigen doubling time).

DETAILED DESCRIPTION:
This is a pilot phase II, open labeled single center study to assess the efficacy of digoxin on inhibiting PCa progression as measured by PSADT. The participants will take study drug digoxin, which is approved by FDA for the treatment of CHF, 125 or 250 mcg orally daily, titrated to the level of 0.8 - 2 ng/ml for total of 6 cycles (4 weeks/cycle). The lower dose of digoxin (such as 125 mcg/day) will be chosen if serum level reaches 0.8 ng/ml already. Patients may continue another 6 cycles if evident of clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* There must be a confirmed biochemical progression. Biochemical progression is defined as three rises in PSA levels, with each PSA determined at least 4 weeks apart, and each PSA value increase >0.2 ng/ml.
* Baseline PSA must be determined within 4 weeks of study entry. At least 3 PSA values are necessary prior to the study entry to calculate PSA doubling time (PSADT) calculator.
* Men with history of radical prostatectomy are required to have baseline PSA >1 ng/ml. Men treated with primary radiation therapy are required to have baseline PSA>2 ng/ml and greater than 150% rise from postradiation nadir.
* PSA doubling time must be between 6 and 24 months.
* All treatments including intermittent hormonal therapy must have been discontinued for > 6 months prior to study entry.
* No clinical or radiological evidence of distant metastases
* ECOG < 2 and adequate organ function
* Men with history of radical prostatectomy are required to have baseline PSA >1 ng/ml. Men treated with primary radiation therapy are required to have baseline PSA>2 ng/ml and greater than 150% rise from postradiation nadir
* Baseline PSA must be determined within 4 weeks of study entry. At least 3 PSA values are necessary to calculate PSA doubling time via PSADT calculator at: http://www.mskcc.org/mskcc/applications/nomograms/PSADoublingTime.aspx. PSA doubling time must be between 6 and 24 months.
* All previous local modalities of treatment, including radiation and surgery, must have been discontinued at least 8 weeks prior to treatment in this study. Patients may have received prior systemic chemotherapy, hormonal therapy, biologic or vaccine therapy. All systemic treatments must have been discontinued for > 6 months prior to study entry.
* Patients receiving intermittent hormonal therapy for their rising PSA state are considered eligible if testosterone level is above 150ng/dl and treatment was discontinued > 6 months and agree not to have additional injections while on study drug.
* No clinical or radiological evidence of distant metastases (excluding prostascint scan/PET in absence of radiographic disease in Bone scan, CT scan or MRI if used). Lymph node up to 2 cm size is allowed for the study.
* ECOG < 2 or Karnofsky Performance status >70% within 14 days before being registered for protocol therapy (Appendix B)
* Normal organ function with acceptable initial laboratory values:
* Absolute neutrophil count ≥ 1 x 109/L
* Platelets > 50 x 109/L
* Creatinine <1.5 mg/dL
* Bilirubin <1.5 X ULN (institutional upper limits of normal)
* AST (SGOT) and ALT (SGPT) ≤ 1.5 x ULN
* Willingness to use adequate methods of contraception throughout study participation and for at least 3 months after completing therapy

Exclusion Criteria:

* Metastatic disease or currently active second malignancy
* History of Sinus Node Disease and AV Block, Accessory AV Pathway (Wolff-Parkinson-White Syndrome), history of Acute Myocardial Infarction.
* Electrolyte imbalance (hypokalemia, hypo- or hypercalcemia, hypomagnesemia)
* Severe pulmonary disease and hypoxia
* Medical conditions such as uncontrolled hypertension, uncontrolled diabetes mellitus, active infectious hepatitis, type A, B or C, hypothyroidism or hyperthyroidism, which would, in the opinion of the investigator, make this protocol unreasonably hazardous.
* Major thoracic or abdominal surgery within the prior 3 weeks.
* Patients with GI tract disease resulting in an inability to take oral medication, malabsorption syndrome, a requirement for IV alimentation, prior surgical procedures affecting absorption, uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis).
* Use of any prohibited concomitant medications: The washout period is at least 2 weeks before starting the study.
* Insufficient time from last prior regimen or radiation exposure: Systemic therapies for prostate cancer within 28 days prior to digoxin; strontium-89 within 12 weeks; bicalutamide within 6 weeks.
* Persistent Grade >2 treatment-related toxicity from prior therapy
* History of any digoxin-related or drug induced anaphylactic reaction
* Receipt of another investigational agent within 6 months of study entry. Patient must have recovered from all side effects of prior investigational therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jianqing Lin, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Digoxin: Patients receive digoxin PO daily. Treatment repeats every 28 days for up to 6-12 courses in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Digoxin
Started | 16
Completed | 13
Not Completed | 3
Not completed — Withdrawal by Subject | 1
Not completed — Severe back pain | 1
Not completed — Ineligible | 1

BASELINE CHARACTERISTICS:
Arm/Group | Digoxin
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.5)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Rate of Positive PSADT Outcome
Description: Proportion of patients at 6 months post-treatment with a PSADT >= 200% from baseline
Time Frame: 6 months after treatment with digoxin
Measure: Number; unit: participants
Arm/Group | Digoxin
Number analyzed (Participants) | 13
participants | 5

ADVERSE EVENTS:
Arm/Group | Digoxin
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Digoxin (N=16)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Change in taste (General disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 2 (4)
Hyperglycemia (Blood and lymphatic system disorders) | 3 (6)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (2)
Hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
Incontinence (General disorders) | 1 (1)
Decreased appetite (General disorders) | 2 (3)
Cold/cough (General disorders) | 3 (3)
Testicular soreness (Reproductive system and breast disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (4)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1)
ALT high (Hepatobiliary disorders) | 2 (3)
Fatigue (General disorders) | 3 (3)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 1 (2)
Bicarbonate low (Blood and lymphatic system disorders) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 2 (2)
Loose stools (General disorders) | 2 (2)
Decreased energy (General disorders) | 1 (1)
Lightheadedness (General disorders) | 2 (2)
Neck pain (General disorders) | 2 (2)
Arm pain (General disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Foot pain (General disorders) | 1 (1)
Numbness/cramping of lower legs (General disorders) | 1 (1)
Abdominal pain (General disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Nausea (General disorders) | 2 (2)
Hypertension (Blood and lymphatic system disorders) | 2 (3)
Headaches (General disorders) | 1 (1)
Back pain (General disorders) | 2 (3)
Vivid dreams (General disorders) | 3 (3)
Nocturia (Renal and urinary disorders) | 1 (1)
Insomnia (General disorders) | 2 (2)
Low libido (General disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Side pain (General disorders) | 1 (1)
Heart palpitations (Cardiac disorders) | 1 (1)
EKG change (Cardiac disorders) | 3 (4)
Rib pain (General disorders) | 1 (1)
Shoulder pain (General disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Tooth root canal (General disorders) | 1 (1)
Difficulty raking deep breaths (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nightmares (General disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Boil on finger (Skin and subcutaneous tissue disorders) | 1 (1)
Acid reflux (Gastrointestinal disorders) | 1 (1)
Knee achiness (Musculoskeletal and connective tissue disorders) | 1 (2)
Poison ivy (Skin and subcutaneous tissue disorders) | 1 (1)
Sinus brachycardia (Cardiac disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes